CLINICAL TRIAL: NCT06385561
Title: The Influence of Tramadol on Opioid-induced Bowel Dysfunction - An Investigator Initiated, Randomized, Double-blinded, Placebo-controlled, Cross-over Clinical Trial
Brief Title: The Influence of Tramadol on Opioid-induced Bowel Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Tramadol_OIBD; 2022-500108-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Opioid-Induced Bowel Dysfunction; Constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Tramadol
  Interventions: Drug: Tramadol
- Placebo treatment (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Tramadol is administered orally twice daily in a dosage of 100 mg (daily total of 200 mg)
  Arms: Active treatment
Drug: Placebo — Placebo is administered orally twice daily.
  Arms: Placebo treatment

SUMMARY:
Tramadol is a weak opioid and widely used to treat moderate to severe pain. Stronger opioids are known to inhibit gastrointestinal motility and secretion, however the effects of tramadol on gastrointestinal function remains less understood. The aim of this study was to determine to what degree tramadol causes opioid-induced bowel dysfunction by using an objective design to explore gastrointestinal transit, motility pattern, secretion, and colonic volume, in a group of healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (assessed by a study-affiliated medical doctor.)
* Signed informed consent.
* Able to read and understand Danish.
* Male (to avoid influence of menstrual cycles)
* Northern European descent (to minimize genetic variance influences on drug metabolism).
* The researcher believes that the participant understands the study details, is compliant and is expected to complete the study.
* Opioid naïve* (who have not taken prescription opioid for one week or longer and at least a year have passed since completion of a previous opioid study.)
* Between 20 and 40 years of age.
* A State Trait Anxiety Inventory (STAI) score in the range of 20-37 i.e., classified as "no or low anxiety" at inclusion.

Exclusion Criteria:

* Known hypersensitivity or allergy towards the used pharmaceutical compounds or pharmaceutical compounds similar to those used in the study.
* Less than three spontaneous bowel movements per week.
* Participation in other studies within 14 days prior to first visit.
* Expected need of medical/surgical treatment during the study.
* Any diagnosed disease, which investigator concludes will affect the trial (including all contraindicated complications: severe chronic obstructive pulmonary disease, pulmonary heart disease, severe bronchial asthma, paralytic ileus, hypercapnia, serious respiratory depression with hypoxia, moderate to severe decreased liver function, gastrointestinal obstruction or perforation, acute surgical abdominal complications such as appendicitis, Mb. Crohn's, ulcerative colitis, and toxic mega colon).
* History of substance abuse (alcohol, tetrahydrocannabinol (THC), benzodiazepine, central stimulants and/or opioids, urine drug test will be performed prior to treatment start). ¹
* History of major mental disorders (e.g., major anxiety, major depression or treatment with psychoactive medications etc.) ²
* Metal implants or pacemaker.
* Daily use of prescription only medicine
* Daily alcohol consumption
* Participation motivated by "wrongful" reasons such as poor economy, or psychosocial issues e.g., problems in the family, loneliness, sadness. People with such problems may be more likely to develop substance dependence.1
* Intake of alcohol within 48 hours before start of study period or any alcohol consumption during each study period. If consumption takes place during the study the participant will be excluded.
* Use of any analgesic medication within 48 hours before start as well as for the duration of the study. If consumption takes place during the study the participant will be excluded.
* Nicotine use

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Total gastrointestinal transit time | From day 4 to day 8
  Difference in hours from ingestion of a 3D Transit Capsule to expulsion of the capsule during active and placebo treatment
Colorectal transit time | From day 4 to day 8
  Difference in hours from the entering in the colon of a 3D Transit Capsule to expulsion of the capsule during active and placebo treatment

SECONDARY OUTCOMES:
Constipation symptoms | From day 1 to day 10
  Measured on the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire (ranging from 0 (symptom absent) to 4 (very severe).
Bowel movement frequency | From day 1 to day 10
  Number of spontaneous bowel movements per day
Stool consistency | From day 1 to day 10
  Rated on the Bristol Stool Form Scale (ranging from type 1 (constipation) - type 7 (diarrhea))
Gastrointestinal symptoms | Day 1 and day 10
  Measured on the Gastrointestinal Symptom Rating Score (GSRS) questionnaire (ranging from 0 (no discomfort) to 6 (very severe discomfort)
Opioid-induced constipation | Day 1 and day 10
  Measured by the Bowel Function Index (BFI) questionnaire (ranging from 0 (not at all) to 100 (very strong).
Diagnostic evaluation of opioid-induced constipation | Day 10
  Assessed using the Rome IV C6 criteria consisting of 7 items rated as either true or false. 2 or more items rated as "true" indicates functional constipation
Colonic motility patterns | From day 4 to day 8
  Number of motility patterns in the colon measured by the 3D Transit Capsule
Opiate withdrawal symptoms | Day 13, 14 or 15
  Measured by the Subjective Opiate Withdrawal Scale (ranging from 0 (not at all) to 4 /extremely)
Colon volume | Day 10
  Volumetric quantification of the colon measured using T2-weighted MRI images
Colonic water content | Day 10
  Analysis of colonic water content measured using heavily T2-weighted MRI images
Gastric half emptying time | Day 1 and day 10
  Analysis of gastric half emptying time after ingestion of a standardized meal measured by MRI
Gastric contraction assessment | Day 1 and day 10
  Analysis of gastric contraction amplitude after ingestion of a standardized meal measured by MRI
Gastric contraction assessment | Day 1 and day 10
  Analysis of gastric contraction frequency after ingestion of a standardized meal measured by MRI
Small bowel motility assessment | Day 1 and day 10
  Analysis of small bowel motility after ingestion of a standardized meal measured using dynamic MRI images. A semi-automated analysis software enables registration of small bowel motility with the calculation of regional motility maps and quantification of motility indices.
Small bowel water content | Day 1 and day 10
  Analysis of small bowel water content measured using heavily T2-weighted MRI images

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be provided upon request